CLINICAL TRIAL: NCT06013800
Title: Volume Status Analysis by Point-of-care Ultrasound: a Cohort Study in Hyponatremia in Internal Medicine
Brief Title: Hyponatremia Volume Status Analysis by Point-of-care Ultrasound
Acronym: Vostaus
Status: Active, not recruiting | Type: Observational
Sponsor: Universidad Veracruzana (Other)
Responsible Party: Principal Investigator, Alejandro Martínez Carreón, Principal Investigator, Universidad Veracruzana
Other Study IDs: 01-93-254-2023
Record Dates: First submitted 2023-08-11; First posted 2023-08-28 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Hyponatremia; Water-Electrolyte Imbalance
Keywords: hyponatremia; water-electrolyte imbalance; POCUS; Point-of-care ultrasound
MeSH Terms: conditions — Hyponatremia; Water-Electrolyte Imbalance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Same Volume Status (Clinical and Point-of-Care Ultrasound): The patient has the same volume status clinically and by point-of-care ultrasound
  Interventions: Other: Measurement of sodium levels
- Different Volume Status (Clinical or Point-of-Care Ultrasound): The patient has a different volume status clinically or by point-of-care ultrasound
  Interventions: Other: Measurement of sodium levels

INTERVENTIONS:
Other: Measurement of sodium levels — Patients will get measurements of sodium levels daily in the first 48 hours, then daily or every other day until normal sodium levels (>135mEq/L).

SUMMARY:
This observational study aims to analyze the time of correction of hyponatremia in patients within an internal medicine ward. The researchers will assess volume status using both clinical evaluation and point-of-care ultrasound. Patients will be categorized based on whether they have the same volume status determined clinically and by ultrasound or a different status between the two methods. By tracking sodium levels daily until normalization, the study will compare the time of hyponatremia correction between the two groups.

DETAILED DESCRIPTION:
The main question it aims to answer are What is the time of correction of hyponatremia by assessing the volume status clinically or by point of care of ultrasound?.

Participants will be asked to participate in the study and they will be receive a volume status by a portable ultrasound. If they have the same volume status clinically and by point of care ultrasound they will be referred as group 1. If they have a different volume status clinically or by point of care ultrasound they will be referred as group 2.

Researchers will follow the patients by measuring the sodium levels daily until they reach normal sodium levels ( >135mEq/L) and will compare group 1 and group 2 with a survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years
* Hypotonic hyponatremia (less than 275mosm/kg) calculated by the following formula (2 Na+Glucose/ 18)

Exclusion Criteria:

* Patients who are critically ill with ventilatory support.
* Patients with clinical signs suggestive of hypovolemia and have a documented history of aortic insufficiency or show mitral insufficiency during POCUS (Point-of-Care Ultrasound).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hypotonic hyponatremia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with sodium level >135mEq/L | Baseline, everyday up to 30 days
  Rate of Achieving a Normal Sodium Level (>135mEq/L) per Participant:
  This information will be visually represented through Group 1 and Group 2 using a Kaplan-Meier curve. Subsequently, the data will be evaluated using the Log-Rank test or the Breslow test for statistical significance.

SECONDARY OUTCOMES:
Assessment of clinical variables associated with corrected sodium levels | Baseline, up to 30 days
  To analyze whether the relationship between point-of-care ultrasound-assessed volume status and clinical variables-such as hypertonic saline administration, chronic liver disease, diuretic use, active cancer, type of hospital admission, severity of hyponatremia, and antidepressant use-influences corrected sodium levels.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Martínez Carreón, MD, Principal Investigator — Universidad Veracruzana
Locations (1):
- Hospital Regional B Veracruz Alta Especialidad, Veracruz, Mexico